CLINICAL TRIAL: NCT06161467
Title: Transcutaneous Laryngeal Ultrasoungraphy (TLUS) as an Alternative to Direct Flexible Laryngoscopy (DFL) in Assessment of Vocal Cords Appearance in Patients Underwent Thyroid Surgery
Brief Title: Transcutaneous Laryngeal Ultrasound as an Alternative to Direct Flexible Laryngoscopy in Assessment of Vocal Cords
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Mohamed Ali sayd, Principal Investigator, Assiut University
Other Study IDs: vocal cords in US
Record Dates: First submitted 2023-09-19; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Ultrasound Therapy; Complications
Keywords: Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: Ultrasound devices — Safe , no radiation

SUMMARY:
To evaluate the diagnostic value of ultrasound in the assessment of the vocal cords compared with direct flexible laryngoscopy

DETAILED DESCRIPTION:
Thyroid and parathyroid surgery are the most common procedures in endocrine surgery worldwide. They are mainly associated with two major complications: recurrent laryngeal nerve (RLN) palsy and hypoparathyroidism, The preservation of recurrent laryngeal nerve (RLN) is an essential part of thyroid surgery {1}. The various methods to test the normal functionality of vocal cords (VCs) include direct visualisation under the fiber bronchoscope, indirect laryngoscopy, laryngeal muscles electromyography, computed tomography (CT), and magnetic resonance imaging (MRI). We aimed to assess the usefulness of ultrasound (USG) in the examination of VC morphology and movement.

Recurrent laryngeal nerve injury ranges from 1.4 to 5.1% following surgery involving the thyroid gland.

Otolaryngology and Head and Neck Surgery suggested that all patients undergoing thyroid and parathyroid procedures should undergo routinely preoperative and postoperative DFL [6].

Laryngoscopy is considered the golden standard to evaluate vocal fold mobility preoperatively. As it can demonstrate a paralysis of the recurrent laryngeal nerve,. Yet it is not common practice for many endocrine surgery teams because it is time consuming, imposes extra costs, and is in general, an unpleasant experience for some patients.{2} head and neck ultrasonography is a cost effective imaging tool that is currently used as an extension of patient physical examination. That is based on its safety (non invasive and non ionizing radiation dependent), repeatability, availability and good patient compliance (pain less and require no sedation). {3} recently portable ultrasound devices became widely available with dramatic improvement of the imaging quality rendering to increased diagnostic accuracy. Availability, usability and mobility of the devices encourage bedside examination which is essential in non mobile patient and ICU patient [4] .

However, the experience is limited and the reliability of the TLUS in thyroid and parathyroid surgery is still being debated

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thyroid surgery
* Patients underwent thyroid surgery

Exclusion Criteria:

• Patients with vocal cord paralysis because of any cause other than thyroid surgery complications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Vocal cords appearance | Two years
  Assessment of vocal cords appearance by Transcutaneous laryngeal ultrasoungraphy (TLUS) as an alternative to direct flexible laryngoscopy (DFL)
Vocal cords movement | Two years
  Assessment of vocal cords movement by Transcutaneous laryngeal ultrasoungraphy (TLUS) as an alternative to direct flexible laryngoscopy (DFL)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Farouk, Professor, Principal Investigator — Supervisor

REFERENCES:
- [Background] American Thyroid Association (ATA) Guidelines Taskforce on Thyroid Nodules and Differentiated Thyroid Cancer; Cooper DS, Doherty GM, Haugen BR, Kloos RT, Lee SL, Mandel SJ, Mazzaferri EL, McIver B, Pacini F, Schlumberger M, Sherman SI, Steward DL, Tuttle RM. Revised American Thyroid Association management guidelines for patients with thyroid nodules and differentiated thyroid cancer. Thyroid. 2009 Nov;19(11):1167-214. doi: 10.1089/thy.2009.0110. PMID 19860577
- [Background] Holtel MR. Emerging technology in head and neck ultrasonography. Otolaryngol Clin North Am. 2010 Dec;43(6):1267-74, vii. doi: 10.1016/j.otc.2010.08.003. PMID 21044741